CLINICAL TRIAL: NCT06775119
Title: Feasibility Study of a Neuromuscular Fatigue Test and Associated Hemodynamic Responses: Application in Healthy Volunteers for Use in Patients with Chemotherapy-treated Breast Cancer
Acronym: PROTECT-08A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-002
Record Dates: First submitted 2024-08-12; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Fatigue; Muscle; Heart
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental protocol (Experimental)
  Interventions: Other: Test of neuromuscular fatigue and associated hemodynamic responses

INTERVENTIONS:
Other: Test of neuromuscular fatigue and associated hemodynamic responses — Baseline measurements of neuromuscular function and hemodynamic responses will be done. Investigators will then assess the mechanoreflex activation using the experimental technique of passive leg movement (PLM).
  Following the PLM and the neuromuscular function baseline assessments, participants will perform four consecutive blocks, each consisting of a fatigue task followed by post-exercise circulatory occlusion (PECO). Neuromuscular function, assessed through maximal voluntary contraction (MVC) and quadriceps twitch techniques, will be measured before the fatigue task and after PECO in each block. Participants will perform 2-minutes isometric quadriceps sustained contraction at 20% MVC to induce exercise-induced neuromuscular fatigue. Hemodynamic responses will be measured during the PECO to isolate to the metaboreflex by inflating a cuff over the right thigh for a 2 minutes duration. After the PECO, the thigh cuff will be deflated, and neuromuscular function will be reassessed.

SUMMARY:
This cross-sectional and single-center study aims to progressively induce an increase in peripheral fatigue during successive efforts in healthy subjects. Participants will undergo three evaluations, each lasting one and half hours, to validate the test and assess its reproducibility. These three visits will be conducted at a minimum interval of 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* Informed consent
* Age ≥ 18 years old
* Affiliation to a social security system
* Able to speak, read and understand French
* Practice physical activity 1 to 5 times per week, without reaching a level of intense training or high-level performance.

Exclusion Criteria:

* History of cancer
* Any known chronic pathology
* Protected minor or adult
* Psychiatric, musculoskeletal or neurological problems
* Implantation of a pacemaker
* Pregnant woman
* Presenting at least one contraindication to the use of transient blood flow occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of the progressive changes in the level of peripheral fatigue through the consecutive blocks. | All measurements will be taken at the end of each of the four exercise bouts, during the same visit.
  Significant changes in the level of peripheral fatigue during successive efforts as measured by the non invasive technique of nervous stimulation of the motor nerve.

SECONDARY OUTCOMES:
Correlation between peripheral fatigue and haemodynamic responses | Correlation between variables measured at the end of each of the four exercise bouts, during the same visit
  Correlation between the level of change in the amplitude of the potentiated quadriceps twitch and the level of change in haemodynamic parameters.
Validate the feasibility of the test on the following secondary parameter: reproducibility of the test | 2 to 7 days between sessions 2 and 3.
  Reproducibility of the test due to the absence of significant difference in the exercise-induced peripheral fatigue levels (percentage change from baseline) and mean arterial pressure (mmHg) between sessions 2 and 3.
Validate the feasibility of the test on the following secondary parameter: absence of transient discomfort | All measurements will be taken at the end of each of the four exercise bouts, during the same visit
  Low rating of the level of discomfort assessed by a 10 cm visual analog scale after each effort. The participant will be asked to grade between 0 and 10 the level of discomfort felt in the thighs.
Validate the feasibility of the test on the following secondary parameter: Tolerance to peripheral nerve stimulation using the self-reports of pain intensity scales. | All measurements will be taken during the same visit, at the end of each of the four exercise bouts
  Evaluation of the subject's response to various levels of peripheral nerve stimulation intensity, starting with very low intensities, while recording any sensations of discomfort reported by the subject using the self-reports of pain intensity scales (10 cm visual analog scale).

CONTACTS AND LOCATIONS:
Overall Officials: Roland SCHOTT, MD, Principal Investigator — Institut de cancérologie Strasbourg Europe
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France